CLINICAL TRIAL: NCT04904588
Title: A Multi-Center, Phase II Trial of HLA-Mismatched Unrelated Donor Hematopoietic Cell Transplantation With Post-Transplantation Cyclophosphamide for Patients With Hematologic Malignancies
Brief Title: HLA-Mismatched Unrelated Donor Hematopoietic Cell Transplantation With Post-Transplantation Cyclophosphamide
Acronym: ACCESS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCESS
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Mixed Phenotype Acute Leukemia; Acute Leukemia; Myelodysplastic Syndromes; Chronic Myelogenous Leukemia; Chronic Lymphocytic Leukemia; Lymphoma
Keywords: Lymphoma; Leukemia; Hematologic Diseases; Myelodysplastic Syndromes; Preleukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Bone Marrow Diseases; Precancerous Conditions; Leukemia, Lymphoid; Leukemia, B-Cell; Leukemia, Myeloid; Cyclophosphamide; Mesna; Tacrolimus; Busulfan; Fludarabine; Total Body Irradiation; Melphalan; Mycophenolate mofetil; Immunosuppressive Agents; Immunologic Factors; Physiological Effects of Drugs; Hematopoietic Stem Cell Transplantation; Unrelated Donors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Leukemia; Hematologic Diseases; Preleukemia; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Bone Marrow Diseases; Precancerous Conditions; Leukemia, Lymphoid; Leukemia, B-Cell; Leukemia, Myeloid | interventions — Busulfan; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Cyclophosphamide; Melphalan; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation; Mesna; Tacrolimus; Mycophenolic Acid; Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Regimen A (MAC: busulfan and fludarabine, PBSC HCT) (Experimental): Patients receive:
  * Busulfan (≥ 9 mg/kg total dose) IV or PO on days -6 to -3
  * Fludarabine (150 mg/m2 total dose) IV on days -6 to -2
  Patients receive a peripheral blood stem cell (PBSC) graft infusion from a mismatched unrelated donor on Day 0.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-transplant Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient-Reported Outcomes
- Regimen B (MAC: Fludarabine and TBI; PBSC HCT) (Experimental): Patients receive:
  * Fludarabine (90 mg/m2 total dose) IV on days -7 to -5
  * Total body irradiation (TBI) (1200 cGy total dose) on days -4 to -1
  Patients receive a PBSC graft infusion from a mismatched unrelated donor on Day 0.
  Interventions: Drug: Fludarabine; Radiation: Total-body irradiation; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-transplant Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient-Reported Outcomes
- Regimen C (RIC: Fludarabine and Busulfan; PBSC HCT) (Experimental): Patients receive:
  * Fludarabine (120-180 mg/m2 total dose) IV on days -6 to -2
  * Busulfan (less than or equal to 8 mg/kg PO or 6.4 mg/kg IV) on days -5 and -4
  Patients receive a PBSC graft infusion from a mismatched unrelated donor on Day 0.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-transplant Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient-Reported Outcomes
- Regimen D (RIC: Fludarabine and Melphalan; PBSC HCT) (Experimental): Patients receive:
  * Fludarabine (120-180 mg/m2 total dose) IV on days -7 to -3
  * Melphalan (100-140 mg/m2) IV on day -1
  Patients receive a PBSC graft infusion from a mismatched unrelated donor on Day 0.
  Interventions: Drug: Fludarabine; Drug: Melphalan; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-transplant Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient-Reported Outcomes
- Regimen E (NMA: Fludarabine, Cyclophosphamide, TBI; PBSC HCT) (Experimental): Patients receive:
  * Fludarabine (150 mg/m2 total dose) IV on days -6 to -2
  * Cyclophosphamide (29-50 mg/kg) IV on days -6 and -5
  * TBI (200 cGy) on day -1
  Patients receive a PBSC graft infusion from a mismatched unrelated donor on Day 0.
  Interventions: Drug: Fludarabine; Radiation: Total-body irradiation; Drug: Cyclophosphamide; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-transplant Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient-Reported Outcomes
- Regimen F (MAC: Busulfan and Cyclophosphamide; BM HCT) (Experimental): Patients receive:
  * Busulfan (dosed by age and weight per institutional standards to target goal pharmacokinetic (PK) in range noted in protocol.) on days -6 to -3
  * Cyclophosphamide (100 mg/kg total dose) IV on days -2 and -1
  Patients receive a bone marrow (BM) graft infusion from a mismatched unrelated donor on Day 0.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Procedure: Bone Marrow Hematopoietic Stem Cell Transplantation; Drug: Post-transplant Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient-Reported Outcomes
- Regimen G (MAC: Cyclophosphamide and TBI; BM HCT) (Experimental): Patients receive:
  * Cyclophosphamide (100 mg/kg total dose) IV on days -5 and -4
  * TBI (1200 cGy total dose) on days -3, -2 and -1
  Patients receive a BM graft infusion from a mismatched unrelated donor on Day 0.
  Interventions: Radiation: Total-body irradiation; Drug: Cyclophosphamide; Procedure: Bone Marrow Hematopoietic Stem Cell Transplantation; Drug: Post-transplant Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient-Reported Outcomes

INTERVENTIONS:
Drug: Busulfan — Given IV or PO pre-transplant as part of conditioning regimen
  Other Names: Busulfex®
  Arms: Regimen A (MAC: busulfan and fludarabine, PBSC HCT); Regimen C (RIC: Fludarabine and Busulfan; PBSC HCT)
Drug: Busulfan — Given IV pre-transplant as part of conditioning regimen
  Other Names: Busulfex®
  Arms: Regimen F (MAC: Busulfan and Cyclophosphamide; BM HCT)
Drug: Fludarabine — Given IV pre-transplant as part of conditioning regimen
  Other Names: Fludara®
  Arms: Regimen A (MAC: busulfan and fludarabine, PBSC HCT); Regimen B (MAC: Fludarabine and TBI; PBSC HCT); Regimen C (RIC: Fludarabine and Busulfan; PBSC HCT); Regimen D (RIC: Fludarabine and Melphalan; PBSC HCT); Regimen E (NMA: Fludarabine, Cyclophosphamide, TBI; PBSC HCT)
Radiation: Total-body irradiation — Administered pre-transplant as part of conditioning regimen
  Other Names: TBI
  Arms: Regimen B (MAC: Fludarabine and TBI; PBSC HCT); Regimen E (NMA: Fludarabine, Cyclophosphamide, TBI; PBSC HCT); Regimen G (MAC: Cyclophosphamide and TBI; BM HCT)
Drug: Cyclophosphamide — Given IV pre-transplant as part of conditioning regimen
  Other Names: Cytoxan®
  Arms: Regimen E (NMA: Fludarabine, Cyclophosphamide, TBI; PBSC HCT); Regimen F (MAC: Busulfan and Cyclophosphamide; BM HCT); Regimen G (MAC: Cyclophosphamide and TBI; BM HCT)
Drug: Melphalan — Given IV pre-transplant as part of conditioning regimen
  Arms: Regimen D (RIC: Fludarabine and Melphalan; PBSC HCT)
Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT) — Peripheral blood stem cell graft is infused from a mismatched unrelated donor on Day 0.
  Other Names: PBSC HSCT; PBSC HCT; PBSC Transplantation
  Arms: Regimen A (MAC: busulfan and fludarabine, PBSC HCT); Regimen B (MAC: Fludarabine and TBI; PBSC HCT); Regimen C (RIC: Fludarabine and Busulfan; PBSC HCT); Regimen D (RIC: Fludarabine and Melphalan; PBSC HCT); Regimen E (NMA: Fludarabine, Cyclophosphamide, TBI; PBSC HCT)
Procedure: Bone Marrow Hematopoietic Stem Cell Transplantation — Bone marrow graft is infused from a mismatched unrelated donor on Day 0.
  Other Names: BM HSCT; BM HCT; Bone Marrow Transplantation
  Arms: Regimen F (MAC: Busulfan and Cyclophosphamide; BM HCT); Regimen G (MAC: Cyclophosphamide and TBI; BM HCT)
Drug: Post-transplant Cyclophosphamide — Cyclophosphamide (50 mg/kg) is administered on Day +3 and on Day +4 post-transplant as an IV infusion over 1-2 hours.
  Other Names: Cytoxan®
Drug: Mesna — Mesna is given in divided doses IV 30 min pre- and at 3, 6, and 8 hours post-cyclophosphamide.
  Other Names: Mesnex®
Drug: Tacrolimus — Tacrolimus is given at a dose of 0.05 mg/kg PO or an IV dose of 0.03 mg/kg of ideal body weight (IBW) starting on Day +5 post-transplant with taper recommended at 90-100 days post HCT.
Drug: Mycophenolate Mofetil — Mycophenolate mofetil (MMF) is given at a dose of 15 mg/kg three times daily IV or PO from Day +5 to Day +35 post-transplant.
  Other Names: MMF; Cellcept®
Other: Patient-Reported Outcomes — Survey assessments will be administered to study participants pre- and post-transplant.

SUMMARY:
This is a prospective, multi-center, Phase II study of hematopoietic cell transplantation (HCT) using human leukocyte antigen (HLA)-mismatched unrelated donors (MMUD) for peripheral blood stem cell transplant in adults and bone marrow stem cell transplant in children. Post-transplant cyclophosphamide (PTCy), tacrolimus and mycophenolate mofetil (MMF) will be used for for graft versus host disease (GVHD) prophylaxis. This trial will study how well this treatment works in patients with hematologic malignancies.

ELIGIBILITY:
Stratum 1 Recipient Inclusion Criteria:

1. Age > 18 years and < 66 years (chemotherapy-based conditioning) or < 61 years (total body irradiation [TBI]-based conditioning) at the time of signing informed consent
2. Planned MAC regimen as defined per protocol
3. Available partially HLA-MMUD (4/8-7/8 at HLA-A, -B, -C, and -DRB1 is required) with age < 35 years
4. Product planned for infusion is PBSC
5. HCT Comorbidity Index (HCT-CI) < 5
6. One of the following diagnoses:

   1. Acute myeloid leukemia (AML) acute lymphoblastic leukemia (ALL), or other acute leukemia in 1st remission or beyond with ≤ 5% marrow blasts and no circulating blasts or evidence of extra-medullary disease. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   2. Patients with myelodysplastic syndrome (MDS) with no circulating blasts and with < 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with < 5% or 5-10% blasts in MDS). Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
7. Cardiac function: Left ventricular ejection fraction > 45% based on most recent echocardiogram or multigated acquisition scan (MUGA) results
8. Estimated creatinine clearance > 60 mL/min calculated by equation
9. Pulmonary function: diffusing capacity of the lungs for carbon monoxide (DLCO) corrected for hemoglobin > 50% and forced expiratory volume in first second (FEV1) predicted > 50% based on most recent pulmonary function test results
10. Liver function acceptable per local institutional guidelines
11. Karnofsky performance status (KPS) of > 70%
12. Subjects ≥ 18 years of age or legally authorized representative must have the ability to give informed consent according to applicable regulatory and local institutional requirements.

Stratum 2 Recipient Inclusion Criteria

1. Age > 18 years at the time of signing informed consent
2. Planned NMA/RIC regimen as defined per protocol
3. Available partially HLA-MMUD (4/8-7/8 at HLA-A, -B, -C, and -DRB1 is required) with age < 35 years
4. Product planned for infusion is PBSC
5. One of the following diagnoses:

   1. Patients with acute leukemia or chronic myeloid leukemia (CML) with no circulating blasts, no evidence of extramedullary disease, and with < 5% blasts in the bone marrow. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   2. Patients with MDS with no circulating blasts and with < 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with < 5% or 5-10% blasts in MDS.) Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   3. Patients with chronic lymphocytic leukemia (CLL) or other leukemias (including prolymphocytic leukemia) with chemosensitive disease at time of transplantation
   4. Patients with lymphoma with chemosensitive disease at the time of transplantation
6. Cardiac function: Left ventricular ejection fraction > 45% based on most recent echocardiogram or MUGA results with no clinical evidence of heart failure
7. Estimated creatinine clearance > 60 mL/min calculated by equation
8. Pulmonary function: DLCO corrected for hemoglobin > 50% and FEV1 predicted > 50% based on most recent pulmonary function test results
9. Liver function acceptable per local institutional guidelines
10. KPS of > 60%
11. Subjects ≥ 18 years of age or legally authorized representative must have the ability to give informed consent according to applicable regulatory and local institutional requirements.

Stratum 3 Recipient Inclusion Criteria

1. Age > 1 years and < 21 years at the time of signing informed consent
2. Partially HLA-MMUD (4/8-7/8 at HLA-A, -B, -C, and -DRB1 is required) with age < 35 years
3. Product planned for infusion is BM
4. Planned MAC regimen as defined per protocol
5. One of the following diagnosis:

   1. AML in 1st remission or beyond with ≤ 5% marrow blasts, no circulating blasts or evidence of extra-medullary disease. Pre-transplant MRD testing will be performed as per standard of practice at the treating institution. Patients with any MRD status are eligible and should be enrolled at the discretion of provider. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   2. Patients MDS with no circulating blasts and less than 10% blasts in the bone marrow. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   3. ALL in 1st remission or beyond with ≤ 5% marrow blasts, no circulating blasts, or evidence of extra-medullary disease. Pre-transplant MRD testing will be performed as standard practice at the treating institution with the goal of achieving MRD of <0.01%. Patients with any MRD status are eligible and should be enrolled at the discretion of provider. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   4. Other leukemia (mixed-phenotype acute leukemia [MPAL], CML, or other leukemia) in morphologic remission with ≤ 5% marrow blasts and no circulating blasts or evidence of extramedullary disease. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   5. Chemotherapy sensitive lymphoma in at least partial remission (PR)
6. KPS or Lansky performance score ≥ 70%
7. Cardiac function: Left ventricular ejection fraction of ≥ 50% and shortening fraction of ≥ 27% based on most recent echocardiogram
8. Glomerular Filtration Rate (GFR) of ≥ 60ml/min/1.73m2 measured by nuclear medicine scan or calculated from a 24 hour urine collection
9. Pulmonary function: DLCO corrected for hemoglobin, FEV1, and Forced Vital Capacity (FVC) of ≥50% if able to perform pulmonary function tests. If unable to perform pulmonary function tests, must have a resting pulse oximetry of >92% without supplemental oxygen.
10. Hepatic: Total bilirubin ≤ 2.5 mg/dL and alanine aminotransferase (ALT), aspartate aminotransferase (AST) < 3x the upper limit of normal
11. Legal guardian permission must be obtained for subjects < 18 years of age. Pediatric subjects will be included in age appropriate discussion in order to obtain assent.
12. Subjects ≥ 18 years of age or legally authorized representative must have the ability to give informed consent according to applicable regulatory and local institutional requirements.

Donor Inclusion Criteria:

1. Must be unrelated to the subject and high-resolution HLA-matched at 4/8, 5/8, 6/8, or 7/8 (HLA-A, -B, -C, and -DRB1)
2. Donor must be typed at high-resolution for a minimum of HLA-A, -B, -C, -DRB1, -DQB1, and -DPB1
3. Age > 18 years and < 35 years at the time of signing informed consent
4. Meet the donor registries' medical suitability requirements for PBSC or BM donation
5. Must undergo eligibility screening according to current Food and Drug Administration (FDA) requirements. Donors who do not meet one or more of the donor screening requirements may donate under urgent medical need.
6. Must agree to donate PBSC (or BM for stratum 3)
7. Must have the ability to give standard (non-study) informed consent according to applicable donor regulatory requirements

Recipient Exclusion Criteria (Strata 1, 2 and 3):

1. Suitable HLA-matched related or 8/8 high-resolution matched unrelated donor available
2. Subject unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
3. Primary myelofibrosis or myelofibrosis secondary to essential thrombocythemia, polycythemia vera, or MDS with grade 4 marrow fibrosis
4. Subjects with a prior allogeneic HSC transplant
5. Subjects with an autologous HSC transplant within the past 3 months
6. Females who are breast-feeding or pregnant
7. Uncontrolled bacterial, viral or fungal infection at the time of the transplant preparative regimen
8. Concurrent enrollment on other interventional GVHD clinical trial (enrollment on supportive care trials may be allowed after discussion with Principal Investigators)
9. Subjects who undergo desensitization to reduce anti-donor HLA antibody levels prior to transplant.
10. Patients who are HIV+ with persistently positive viral load. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.

Donor Exclusion Criteria:

1. Donor unwilling or unable to donate
2. Recipient positive anti-donor HLA antibodies against a mismatched HLA in the selected donor determined by the presence of donor specific HLA antibodies (DSA) to any mismatched HLA allele/antigen at any of the following loci (HLA-A, -B, -C, -DRB1, DRB3, DRB4, DRB5, -DQA1, -DQB1, -DPA1, -DPB1) with median fluorescence intensity (MFI) >3000 by microarray-based single antigen bead testing. In patients receiving red blood cell or platelet transfusions, DSA evaluation must be performed or repeated post-transfusion and prior to donor mobilization and initiation of recipient preparative regimen.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 year post HCT

SECONDARY OUTCOMES:
Event-free survival | 1 year post-HCT
  Defined as graft failure, relapse or progression of underlying disease, death, grade 3-4 acute GVHD, or NIH-severe chronic GVHD.
GVHD, relapse free survival | 1 year post-HCT
  Defined as relapse or progression of underling disease, graft failure, grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, or death by any cause.
Modified GVHD, relapse free survival | 1 year post-HCT
  Defined as relapse or progression of underling disease, graft failure, grade III-IV acute GVHD, NIH moderate or severe chronic GVHD, or death by any cause.
Progression-free survival | 1 year post-HCT
Cumulative incidence of nonrelapse mortality | Day +100 and 1 year post-HCT
Event-Free Survival based on donor HLA match grade and donor age (7/8 versus <7/8) | 1 year post-HCT
Overall Survival based on donor HLA match grade and donor age (7/8 versus <7/8) | 1 year post-HCT
Cumulative incidence of neutrophil recovery | Day +100 post-HCT
  Defined as neutrophil count ≥500/mm^3 for 3 consecutive days post-HCT.
Kinetics of neutrophil recovery | Day +100 post-HCT
  Defined as the evaluation of the time it takes for neutrophil count recovery to occur in the study subjects.
Cumulative incidence of platelet recovery | Day +100 post-HCT
  Defined as platelet count ≥20,000/mm^3 or ≥50,000/mm^3 with no platelet transfusions within seven days.
Kinetics of platelet recovery | Day +100 post-HCT
  Defined as the evaluation of the time it takes for platelet count recovery to occur in the study subjects.
Cumulative incidence of primary graft failure | Day +28 post-HCT
Donor chimerism | Day +100 post-HCT
  Strata 2 and 3 only. Percent of donor chimerism via peripheral blood
Cumulative incidence of acute GVHD | Day +100 post-HCT
Cumulative incidence of chronic GVHD | 1 year post-HCT
Cumulative incidence of BK and cytomegalovirus (CMV) viral infections | Days +100 and +180 post-HCT
Cumulative incidence of relapse/progression | 1 year post-HCT
Incidence of cytokine release syndrome (CRS) | Day +14 post-HCT
  Overall incidence of CRS of any grade and grade 3 or 4 CRS post-transplant
Cumulative incidence of secondary graft failure | 1 year post-HCT
Overall Toxicity | 1 year post-HCT
  To tabulate adverse events (AEs) experienced by recipients, defined as grade 3-5 unexpected and Grade 5 expected AEs, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Devine, MD, Principal Investigator — NMDP/Be The Match
Locations (39):
- United States (39):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University Medical Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Medical Center - Mott Children's Hospita, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Ohio State Medical Center, James Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - TriStar BMT, Nashville, Tennessee
  - TriStar Medical Group Children's Specialists, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - -Baylor College of Medicine - Texas Children's Hospital and Houston Methodist, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin Hospital and Clinic, Madison, Wisconsin
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Malki MM, Bo-Subait S, Logan B, Olson J, Kou J, Smith S, Leckrone E, Wu J, Stefanski HE, Auletta JJ, Spellman SR, Malmberg C, Askar M, Cusatis R, Shaffer BC, Modi D, Khimani F, Gooptu M, Hamadani M, Madbouly A, Maiers M, Fingerson S, Cook R, Ballen K, Loren A, Larkin K, Arai S, Qayed M, Choi SW, Broglie L, Shaw BE, Devine SM, Jimenez Jimenez AM. Post-Transplant Cyclophosphamide-Based Graft-Versus-Host Disease Prophylaxis After Mismatched Unrelated Donor Peripheral Blood Stem Cell Transplantation. J Clin Oncol. 2025 Sep;43(25):2772-2781. doi: 10.1200/JCO-25-00856. Epub 2025 Jun 16. PMID 40523209